CLINICAL TRIAL: NCT01928342
Title: The Effects of Coenzyme A Combined With Statin on Serum Lipids in Patients With Hyperlipidemia: a Randomized, Double-blinded, Placebo-controlled, Multi-center Clinical Trial
Brief Title: The Effects of Coenzyme A Combined With Statin on Serum Lipids in Patients With Hyperlipidemia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Jiangtao Lai, MD, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012MMXX2CoA008
Record Dates: First submitted 2013-08-16; First posted 2013-08-23 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Hyperlipoproteinemia
MeSH Terms: conditions — Hyperlipoproteinemias | interventions — Coenzyme A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coenzyme A 400mg (Experimental): Coenzyme A 400mg per day
  Interventions: Drug: Coenzyme A
- Placebo (Placebo Comparator): Capsule without coenzyme A.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Coenzyme A — Coenzyme A 400mg per day
  Other Names: Coenzyme A group
  Arms: Coenzyme A 400mg
Drug: Placebo — Capsule without coenzyme A.
  Other Names: Controls.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the lipid lowering effects and clinical safety of a natural hypolipidemic compound, coenzyme A （CoA） capsule, combined use with statin, in Chinese patients with moderate dyslipidemia.

DETAILED DESCRIPTION:
Although lowering cholesterol and low-density lipoprotein-cholesterol (LDL-C) is the mainstay of medical therapy for cardiovascular event prevention, evidence from clinical trials supports a role for elevated triglyceride (TG) and low high-density lipoprotein cholesterol (HDL-C) concentrations in the residual cardiovascular risk on statin treatment. Fenofibrate is the most commonly used agent to control hypertriglyceridemia as monotherapy or combining with statin, which lowers TG and raises HDL-C through multifaceted mechanism by PPARα activation. However, safety of coadministration of statin with fenofibrate has been a great concern, especially drug-induced hepatotoxicity when they are combined used. Coenzyme A (CoA) functions as an acyl group carrier and assists in transferring fatty acids from the cytoplasm to mitochondria. It is also involved in the oxidation and catabolism of fatty acids. Animal studies have proved its lipid-lowering effects. In a previous multicenter study we conducted in 2008, it was found that oral CoA 400U/d effectively lowered serum TG levels in hypertriglyceridemia patients without increasing adverse effects when compared with placebo. So, the present study was performed to further investigate the lipid-lowing effects and safety of CoA capsule combined with statin in dyslipidemia patients.

ELIGIBILITY:
Inclusion Criteria:

* TG 2.3～7.0mmol/l
* 18-80 years of age
* combined use with statins

Exclusion Criteria:

* pregnancy
* acute liver disease or hepatic dysfunction, as determined by levels of alanine aminotransferase (ALT) or aspartate aminotransferase levels (AST) more than 2-fold the upper normal limit
* nephrotic syndrome or serum creatinine (Cr) ≥2-fold the upper normal limit and creatine phosphokinase (CK) more than 3-fold the upper normal limit
* primary hypothyroidism
* psychiatric patients
* poorly controlled hypertension, as indicated by a Systolic Blood Pressure >180 mmHg or Diastolic Blood Pressure >110 mmHg
* using contraceptive agent
* using immunosuppressive drugs, prohibited medication or other non-statin lipid-lowing drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-09 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
serum triglyceride level | 8 weeks
  The primary efficacy variable was the percentage change in serum lipid level from baseline to 4 and 8 weeks of treatment.

SECONDARY OUTCOMES:
serum total cholesterol level | 8 weeks
  change from baseline to 4 and 8 weeks of treatment in serum total cholesterol level
low-density lipoprotein cholesterol level | 8 weeks
  change from baseline to 4 and 8 weeks of treatment in serum low-density lipoprotein cholesterol level.
serum high-density lipoprotein cholesterol level | 8 weeks
  change from baseline to 4 and 8 weeks of treatment in serum high-density lipoprotein cholesterol level.

CONTACTS AND LOCATIONS:
Overall Officials: Junzhu Chen, Study Chair — Zhejiang University
Locations (1):
- 1st Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Lai J, Wu B, Xuan T, Liu Z, Chen J. Efficacy and tolerability of adding coenzyme A 400 U/d capsule to stable statin therapy for the treatment of patients with mixed dyslipidemia: an 8-week, multicenter, double-blind, randomized, placebo-controlled study. Lipids Health Dis. 2014 Jan 2;13:1. doi: 10.1186/1476-511X-13-1. PMID 24382338